CLINICAL TRIAL: NCT06875882
Title: Evaluating Occupational Stress in Surgeons and Musicians: A Multi-modal Pilot Study Using Wearable EEG, Biomarker Analysis and Validated Questionnaires
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1393; NCI-2025-01927 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-03-10; First posted 2025-03-13 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Occupational Stress
MeSH Terms: conditions — Occupational Stress | interventions — Surgeons

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Occupational Stress: This research study is to learn about occupational stress among surgeons and musicians by integrating psychological assessments, neurophysiological measures, and biomarkers. Researchers want to assess and compare factors associated with occupational stress, among surgeons and musicians, such as changes in stress biomarkers before and after surgery or music performance, anxiety, burnout, demographic factors, and brainwave activity linked to stress. It is hoped the information learned in this study can be used to help promote better health outcomes and enhance the well-being of these workforce members. Participants will undergo saliva sample collections and complete questionnaires before and after the performance or surgery.
  Interventions: Behavioral: Occupational Stress in Surgeons and Musicians
- Optional Procedure: Participants may optionally have a surgery or performance recorded and undergo an EEG while watching the recording. These participants will undergo saliva sample collections and complete questionnaires before and after the EEG recording session.
  Interventions: Behavioral: Occupational Stress in Surgeons and Musicians

INTERVENTIONS:
Behavioral: Occupational Stress in Surgeons and Musicians — Participants will complete 5 questionnaires about participants demographics, burnout rates, and anxiety levels after participants consent to this study. These questionnaires will be sent to participants via email and should take about 15-20 minutes to complete.

SUMMARY:
To learn about occupational stress among surgeons and musicians by integrating psychological assessments, neurophysiological measures, and biomarkers.

DETAILED DESCRIPTION:
Primary Objectives • To assess the change in occupational stress among surgeons and musicians by measuring physiological and psychological stress markers.

Endpoints:

* Changes in salivary cortisol levels (before and after surgeries for surgeons and live public performances for musicians).
* Changes in State-Trait Anxiety Inventory-Short (STAI-S) scores (administered pre- and post-surgery/performance).

SECONDARY OBJECTIVES AND ENDPOINTS

• Assessing and comparing anxiety and burnout, based on the MBI, STAI-T, M-PAS, and SCAT, in surgeons and musicians

Endpoints:

* Baseline levels of anxiety and burnout measured using the MBI, M-PAS, STAI-T, and SCAT.
* Emotional exhaustion, depersonalization, and personal accomplishment from the MBI in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Professional musicians (i.e., those with academic or orchestral appointments) or MD Anderson Neurosurgeons
* For Musicians only: You will have a musical performance within three months of study enrollment.

For Neurosurgeons only: You will perform a surgical procedure within three months of study enrollment.

Exclusion Criteria:

* Individuals who are unable to provide informed consent
* Individuals diagnosed with severe cognitive impairments, severe psychiatric disorders, or hearing or visual impairments that could affect participation
* Individuals previously enrolled in the study
* Non-English-speaking musicians and/or surgeons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Rui, DMA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org